CLINICAL TRIAL: NCT04570735
Title: MRI Biomarkers in Diabetic Kidney Disease
Acronym: MR3T - DKD
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A02750-57
Record Dates: First submitted 2020-09-18; First posted 2020-09-30 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Nephropathies
Keywords: obesity; diabetic nephropathies; biomarkers; metabolites
MeSH Terms: conditions — Diabetic Nephropathies; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- patients with type 2 diabetes and diabetic kidney disease
  Interventions: Diagnostic Test: MRI
- patients with type 2 diabetes and no diabetic kidney disease
  Interventions: Diagnostic Test: MRI
- patients with obesity, no diabetes and no kidney disease
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — MRI

SUMMARY:
Diabetic kidney disease is one of the most severe and frequent complications of diabetes. Few preclinical markers are available apart from plasma creatinine and microalbuminuria. These markers are imperfect (some patients with advanced renal disease do not have an increase in markers) and late. Therefor there is an uncovered need to identify complementary biomarkers. Magnetic Resonance Spectroscopy (MRS) is a Magnetic Resonance Imaging (MRI) technique that allows the physiology and biochemistry of human body tissues to be studied in a non-invasive and non-irradiating manner.

ELIGIBILITY:
Inclusion Criteria:

Common to all 3 category

* Male or female,
* Age≥ 35 years,
* Subject free, with legal protection guardianship or curatorship;
* Enrollment in the French Social Security system;
* Informed consent signed by the patient

Obese patients

* BMI >30 kgm² ;
* With no known diabetes;
* estimated glomerular filtration rate (eGFR) > 60 ml/min/1.73m² and urine albumin-creatinin ratio (ACR) < 3 mg/g

Type 2 diabetic patients without kidney disease

- eGFR > 60 ml/min/1.73m² AND ACR < 3 mg/g,

Type 2 diabetic patients with diabetic kidney disease defined as eGFR 30 to 60 ml/min/1.73m² OR ACR > 30 mg/mmol.

Exclusion Criteria:

Age < 35 years History of kidney transplant Any contraindication to an MRI examination Legal protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, persons residing in a health or social establishment, adults under legal protection and finally patients in emergency situations Pregnant or lactating women, women of childbearing age who do not have effective contraception

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes with or without diabetic kidney disease and patients with obesity and no diabetes
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Correlation between morphometric and functional and metabolic biomarker data obtained by magnetic resonance spectroscopy (MRS) in 3 different patient groups | 1 month

SECONDARY OUTCOMES:
Association between MRS biomarkers and annual glomerural filtration rate slope calculated within 3 previous years | 3 years
Correlation between metabolic MRS biomarkers and urine and plasma metabolites quantification. | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No